CLINICAL TRIAL: NCT04891757
Title: A Phase 1, Multicenter, Open-Label, Dose Escalation Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Clinical Activity of Orally Administered FHD-286, as Monotherapy or Combination Therapy, in Subjects With Advanced Hematologic Malignancies
Brief Title: FHD-286 as Monotherapy or Combination Therapy in Subjects With Advanced Hematologic Malignancies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Foghorn Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FHD-286-C-002
Record Dates: First submitted 2021-05-13; First posted 2021-05-18 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-03

CONDITIONS: Advanced Hematologic Malignancy; Relapsed Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia; Relapsed Myelodysplastic Syndromes; Refractory Myelodysplastic Syndromes; Relapsed Chronic Myelomonocytic Leukemia; Refractory Chronic Myelomonocytic Leukemia
Keywords: AML; Relapsed Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia; MDS; Relapsed Myelodysplastic Syndromes; Refractory Myelodysplastic Syndromes; Phase 1; FHD-286; Foghorn; CMML; Refractory Chronic Myelomonocytic Leukemia; Relapsed Chronic Myelomonocytic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — Cytarabine; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- FHD-286 Monotherapy (Experimental): Closed to Enrollment
  Interventions: Drug: FHD-286
- FHD-286 in Combination with LDAC (Experimental): FHD-286 administered orally + LDAC administered subcutaneously
  Interventions: Drug: FHD-286; Drug: Low Dose Cytarabine
- FHD-286 in Combination with Decitabine (Experimental): FHD-286 administered orally + decitabine administered intravenously (IV)
  Interventions: Drug: FHD-286; Drug: Decitabine

INTERVENTIONS:
Drug: FHD-286 — FHD-286 administered orally
Drug: Low Dose Cytarabine — LDAC administered subcutaneously (SC)
  Other Names: LDAC
  Arms: FHD-286 in Combination with LDAC
Drug: Decitabine — Decitabine administered intravenously
  Arms: FHD-286 in Combination with Decitabine

SUMMARY:
This Phase 1, multicenter, open-label, dose escalation study is designed to assess the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary clinical activity of FHD-286 administered orally as monotherapy or combination therapy, in subjects with advanced hematologic malignancies.

DETAILED DESCRIPTION:
This study is primarily intended to evaluate the safety and tolerability of FHD-286 when administered orally as monotherapy or in combination with either LDAC or decitabine to subjects with R/R AML, R/R MDS, and R/R CMML not in blast crisis. In each arm of the study, successive cohorts of participants will receive increasing oral doses of FHD-286 as a single agent or in combination with LDAC or decitabine to determine the RP2D(s) in this population.

The data from this study in subjects with advanced hematologic malignancies, including safety, tolerability, PK/PD findings, and antitumor activity, will form the basis for subsequent clinical development of FHD-286.

ELIGIBILITY:
Key Inclusion Criteria:

1. Subject must be ≥16 years of age.
2. Subject must:

   * Have a confirmed diagnosis of R/R AML, R/R MDS, or R/R CMML not in blast crisis AND
   * Have received ≤4 prior lines of systemic anticancer therapy for their disease under study; subjects who have received >4 prior lines of systemic anticancer therapy for their disease under study must receive Sponsor approval. AND
   * Be an appropriate candidate for treatment with LDAC (Arm A) or decitabine (Arm B)
3. Subject or their parent or legal guardian (when applicable) must be able to understand and be willing to sign an informed consent and, when applicable, subject must sign an assent form.
4. Subject must be willing and able to comply with scheduled study visits and treatment plans.
5. Subject must be willing to undergo all study procedures unless contraindicated due to medical risk.
6. Subject must have an ECOG PS of ≤2.
7. Subject must have a life expectancy of ≥3 months.
8. Subject must have adequate hepatic function.
9. Subject must have adequate renal function.
10. Subject must have a WBC count ≤20×109/L; treatment with a stable dose of hydroxyurea or other cytoreductive agent (eg, cytarabine) to achieve this count is allowed.
11. Subject must have adequate cardiovascular, respiratory, and immune system function.
12. Subject must agree to abide by dietary and other considerations required during the study.
13. Subject must meet timing requirements with respect to prior therapy and surgery
14. Toxicity related to prior therapy must have returned to Grade ≤2 by CTCAE by approximately 14 days before the start of study treatment or be deemed irreversible and stable by the Investigator. Exceptions include alopecia, neuropathy, appropriately controlled endocrine toxicities, and other well-controlled stable toxicities with discussion with the Sponsor.
15. Female subjects must be:

    * postmenopausal; or
    * permanently sterile, or, if sexually active with male partners, these partners must be azoospermic; or
    * nonpregnant, nonlactating, and, if sexually active with fertile male partners, having agreed to use a highly effective method of contraception
16. Male subjects must have documented azoospermia or, if fertile and sexually active, must agree to use a highly effective method of contraception with their partners of childbearing potential

Key Exclusion Criteria:

1. Subject is unable to provide informed consent and/or to follow protocol requirements.
2. Subject:

   * Has undergone chimeric antigen receptor T cell therapy or HSCT within 60 days of the first dose of study treatment OR
   * Has clinically significant GVHD
3. Subject has evidence (or suspicion) of extramedullary involvement, unless approved by Sponsor.
4. Subject has an immediately life-threatening, severe complication(s) of advanced myeloid malignancy, such as uncontrolled bleeding, pneumonia with hypoxia or shock, and/or disseminated intravascular coagulation.
5. Subject has other malignancy that may interfere with the diagnosis and/or treatment of advanced hematologic malignancies.
6. Subject has active HBV or HCV infections; Subject has known positive HIV antibody results, or AIDS-related illness.
7. Subject has an active severe infection that requires anti-infective therapy or has an unexplained temperature of >38.5°C during screening visits or on their first day of study treatment.
8. Subject has an uncontrolled intercurrent illness.
9. Subject has QTcF >470 msec or other factors that increase the risk of QTc prolongation or arrhythmic events.
10. Subject has any other medical or psychological condition, deemed by the Investigator to be likely to interfere with a subject's ability to sign informed consent/assent, cooperate, or participate in the study.
11. Subject has known allergies or hypersensitivities to:

    * All subjects: components of the FHD-286 formulation
    * Arm A: cytarabine or any of the excipients
    * Arm B: decitabine or any of the excipients
12. Subject is unable to tolerate the administration of oral medication or has GI dysfunction that would preclude adequate absorption, distribution, metabolism, or excretion of FHD-286.
13. Subject is receiving any other anticancer investigational agents. Investigational agents to treat non-cancer indications may be permitted with Sponsor approval.
14. Exclusion Criteria #14 was removed.
15. Subject is on medications classified as:

    * Strong CYP3A inhibitors [Exception: Triazole antifungal agents, including those classified as strong CYP3A inhibitors, are permitted.]
    * Strong CYP3A inducers
    * Sensitive CYP3A substrates with narrow TIs [Stable doses of immunosuppressant medications that are sensitive CYP3A4 substrates may be permitted with Sponsor approval.]
16. Subject is on medications with narrow TIs that are sensitive P-gp or BCRP substrates and are administered orally or on medications classified as strong inhibitors of P-gp or BCRP.
17. Administration of PPIs should be stopped or switched to another ARA 7 days before administration of FHD-286.
18. Subject is requiring clinically significant or increasing doses of systemic steroid therapy or any other systemic immunosuppressive medication. Local or targeted steroid and immunosuppressive therapies are acceptable. Appropriate steroid replacement to manage endocrine toxicities resulting from prior anticancer systemic therapy is permitted.
19. Subject has undergone any prior treatment with a BRG1/BRM inhibitor.
20. Subject is pregnant or breastfeeding or is planning to become pregnant within 1 year of the start of study treatment.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2021-06-14 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of AEs, dose-limiting toxicities (DLTs), serious AEs (SAEs), AEs leading to discontinuation, and adverse events of special interest (AESIs); safety laboratory assessments | Up to 18 months

SECONDARY OUTCOMES:
AML: Complete remission (CR) rate | Up to 18 months
AML: Duration of CR | Up 18 months
AML: CR + CR with partial hematologic recovery (CRh) rate | Up 18 months
AML: Duration of CR + CRh | Up 18 months
AML: Transfusion independence rate | Up 18 months
AML: Event free survival (EFS) | Up 42 months
AML: Overall survival (OS) | Up to 42 months
MDS: CR rate | Up to 18 months
MDS & CMML: Duration of CR | Up to 18 months
MDS & CMML: Partial remission (PR) rate | Up to 18 months
MDS & CMML: Duration of PR | Up to 18 months
MDS & CMML: CR + PR | Up to 18 months
MDS & CMML: Duration of CR + PR | Up to 18 months
MDS & CMML: Hematologic Improvement rate | Up to 18 months
MDS & CMML: EFS | Up to 42 months
MDS: OS | Up to 42 months
PK parameter: Area under the plasma concentration time curve (AUC) | Day 1 and day 8 of cycle 1 (each cycle is 28 days)
Plasma concentration vs. time profiles | Day 1 and day 8 of cycle 1 (each cycle is 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Reilly, MD, Study Director — Foghorn Therapeutics
Locations (5):
- United States (5):
  - City of Hope National Medical Center, Duarte, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Background] DiNardo CD, Fathi AT, Kishtagari A, Bhalla KN, Quintas-Cardama A, Reilly SA, Almon C, Patriquin C, Nabhan S, Healy K, Hickman D, Collins MP, Khalil A, Corrigan D, Zhao T, Piel J, Lyons K, Horrigan K, Schuck V, Martin P, Elliott G, Lahr DL, Bosinger M, D'Aco K, Smolen GA, Hentemann M, Loghavi S, Agresta S, Savona MR, Stein EM. A Phase I Study of FHD-286, a Dual BRG1/BRM (SMARCA4/SMARCA2) Inhibitor, in Patients with Advanced Myeloid Malignancies. Clin Cancer Res. 2025 Jun 13;31(12):2327-2338. doi: 10.1158/1078-0432.CCR-24-3790. PMID 40238563